CLINICAL TRIAL: NCT02822573
Title: A Phase 3 Randomized Placebo Controlled Clinical Trial of Donepezil in Chemotherapy Exposed Breast Cancer Survivors With Cognitive Impairment
Brief Title: Phase 3 Randomized Placebo Controlled Clinical Trial of Donepezil
Acronym: Remember
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00041707; 3UG1CA189824-04S1 (NIH); WF-97116 (Other: NCI); NCI-2016-01050 (Registry Identifier: NCI CTRP Trial ID); IRB00041707 (Other: Wake Forest IRB ID); NCI-2016-01050 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: Cognitive Dysfunction; Memory Impairment
Keywords: Donepezil; Cognition; Breast Cancer
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Breast Neoplasms | interventions — Donepezil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil (Active Comparator): Participants will be asked to take one 5 mg tablet of donepezil daily for 6 weeks followed by two 5 mg tablets daily for 18 weeks. After 24 weeks, participants will begin a 12 week wash-out period.
  Interventions: Drug: Donepezil 5 mg
- Placebo (Placebo Comparator): Participants will be asked to take one tablet of matching placebo daily for 6 weeks followed by two tablets daily for 18 weeks. After 24 weeks, participants will begin a 12 week wash-out period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil 5 mg — Participants will be asked to take one 5 mg tablet of donepezil daily for 6 weeks followed by two 5mg tablets daily for 18 weeks. After 24 weeks, participants will begin a 12 week wash-out period.
  Other Names: Aricept
  Arms: Donepezil
Drug: Placebo — Participants will be asked to take one tablet of matching placebo daily for 6 weeks followed by two tablets daily for 18 weeks. After 24 weeks, participants will begin a 12 week wash-out period.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This study is to compare the safety and effects of donepezil (Aricept) for patients reporting cognitive or memory issues after receiving chemotherapy for breast cancer. Patients will receive either donepezil or placebo for 24 weeks. The primary objective is to see if memory improves with the use of donepezil during the study.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study with 24 weeks of exposure to drug or placebo followed by a 12 week wash-out period. Patients who meet the eligibility criteria will be stratified by age (<50, 50-59, 60-69, ≥70) and randomized to donepezil or placebo with equal probability. A total of 276 patients will be enrolled (138 per arm). We expect an accrual rate of 7-10 participants per month based on our prior feasibility study. We expect the study to be complete within 40 months.

Participants will be asked to take one 5mg tablet of donepezil or one tablet of matching placebo orally once a day for 6 weeks followed by two 5mg tablets (10mg total) of donepezil or two placebo tablets orally once a day for 18 weeks. After 24 weeks, participants will begin a 12 week wash-out period.

Time points for performing study assessments. Participants will be administered the cognitive battery of tests and questionnaires at baseline, week 12, week 24 and week 36. In addition, a single vial of blood will be drawn at baseline for apolipoprotein E (APOE) genotyping and subsequent bioassays (pending supplemental funding).

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old with history of invasive breast cancer
* Must have completed at least 4 cycles of adjuvant/neo-adjuvant cytotoxic chemotherapy between 1 and 5 years prior to registration (Ongoing herceptin or other chronic human epidermal growth factor receptor 2 (HER2) directed therapies are allowed).
* Patients receiving ongoing hormonal therapy for breast cancer must be on the same hormonal agent for at least 3 months prior to study registration and plan to continue for the duration of the study (9 months)
* Use of psychotropic medications (anti-depressants, anxiolytics, sleeping aids, narcotics) is permitted (patient will be asked to list any that have been taken within the last 3 days on the recent medication sheet) if dose is stable over previous 12 weeks. Patients who were previously on one of these psychotropic medications and have subsequently discontinued the drug must have been off the medication for at least 4 weeks prior to enrollment. Patients who have been on a psychotropic medication for at least 12 weeks but have recently switched to a medicine in the same class (for example, switching from one selective serotonin reuptake inhibitor (SSRI) antidepressant to a different SSRI antidepressant) need to be on a stable dose of the new medication for at least 4 weeks prior to enrollment to be eligible.
* Self-reported cognitive problem plus a measured memory deficit (score <7 on single trial of Eligibility Pre-screen Hopkins Verbal Learning Test - Revised (HVLT-R) Form 3).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document.
* Must be able to speak English.
* Patients currently taking a moderate risk corrected QT interval (QTc) prolongation medication (see Appendix A) are allowed if one of the following criteria are met: 1) The moderate risk QTc prolongation medication is stopped. The patient should be off the moderate risk QTc prolongation medication for at least 5 half-lives before starting study drug. 2) Patients that continue using a moderate risk QTc prolongation medication must have a normal QTc interval (≤ 460 milliseconds) on a screening ECG following informed consent and prior to study enrollment. These patients will also be monitored at designated study follow-up visits per Section 7.5 (monitored 3-7 days after initiating study drug, at week 3, and 3-7 days after the study drug dose increase with ECG's to assess the QTc interval; the QTc level must be ≤ 500 milliseconds at these time points in order to continue on the study drug). 3) Moderate risk QTc prolongation medications that are only taken occasionally may be stopped at the discretion of the treating site physician. Patients must be off medication for at least 5 half-lives prior to starting study drug to be eligible.
* Patients currently taking a moderate risk bradycardia-causing agent (see Appendix B) are allowed if one of the following criteria are met: 1) The moderate risk bradycardia-causing agent is stopped. The patient should be off the moderate risk bradycardia-causing agent for at least 5 half-lives before starting study drug. 2) Patients that continue using a moderate risk bradycardia-causing agent must have a resting heart rate ≥ 55 beats per minute at screening following informed consent. These patients' resting heart rate will be monitored 3-7 days after initiating study drug, at week 3, and 3-7 days after the study drug dose increase per Section 7.5. 3) Moderate risk bradycardia-causing agents that are only taken occasionally may be stopped at the discretion of the treating site physician. Patients must be off medication for at least 5 half-lives prior to starting study drug to be eligible.

Exclusion Criteria:

* Evidence or suspected recurrent or metastatic disease.
* Prior brain irradiation is not allowed.
* Planned therapy (surgery, radiation, chemotherapy, or immunotherapy) while on the study for brain and/or extracranial primary/metastatic disease.
* Hypersensitivity to donepezil or piperidine derivatives
* Current use of ceritinib
* Current use of Succinylcholine/Acetylcholinesterase Inhibitors(as listed in Appendix C). For patients who have used these medications, they must not have used them within 4 weeks prior to enrollment.
* Current use of high-risk QTc prolonging medication(s). See Appendix D
* Current use of quinidine or systemic ketoconazole (topical ketoconazole is acceptable to use while on study).
* History of dementia, Alzheimer's disease, multi-infarct dementia or clinically significant Cerebrovascular Accident (history of transient ischemic attack (TIA) is allowed).
* Current use of donepezil, galantamine, rivastigmine, tacrine, memantine, methylphenidate, dextroamphetamine, or any other specific cognition enhancing drug(s). For patients who have used these medications, they must not have used them within 4 weeks prior to pre-screening. Patients who plan to start taking a cognition enhancing drug while on this study are also excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to donepezil. Hypersensitivity to donepezil.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, recent myocardial infarction, cardiac arrhythmia.
* Major medical conditions that affect cognition, traumatic brain injury, multiple sclerosis, acute severe fatigue, chronic fatigue syndrome or fibromyalgia.
* Psychiatric illness/social situations that would limit compliance with study requirements including but not limited to a history of schizophrenia, psychosis or substance abuse.
* Untreated current severe depression. Currently treated depression is permitted if treatment is stable.
* Patients with a resting heart rate less than 55 beats per minute, seizure disorder or peptic ulcer disease (PUD).
* History of congenital long QT syndrome or torsades de pointes.
* Screening QTc of > 460 milliseconds will make the patient ineligible.
* Pregnant women are excluded from this study. Following informed consent, women of child-bearing potential will be screened with a serum or urine pregnancy test within 10 days of enrollment. The effects of donepezil on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because donepezil is known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* It is unknown whether donepezil is excreted in breast milk, for this reason women who are currently breast-feeding are not eligible for this study.
* On another intervention study involving medication at the time of enrollment or during participation in this study. (Exception: Patients will remain eligible for this study if they are also enrolled on the Alliance for Clinical Trials in Oncology study (NCT02927249): Aspirin in Preventing Recurrence of Cancer in Patients with HER2 Negative Stage II-III Breast Cancer After Chemotherapy, Surgery, and/or Radiation Therapy. Studies that involve only blood draws or questionnaires are also permitted.)
* Use of investigational drugs likely to affect cognition within 30 days prior to pre-screening visit.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Rapp, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (278):
- United States (278):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Gaston Hematology and Oncology Associates-Belmont, Belmont, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest National Cancer Institute Community Oncology Research Program (NCORP) Research Base is committed to following the NIH Statement on Sharing Research Data. As of July 2018, the Wake Forest (WF) NCORP Research Base (RB) signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI National Clinical Trials Network (NCTN)/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide.
Time Frame: See NIH Policy
Access Criteria: request using link below
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Rapp SR, Dressler EV, Brown WM, Wade JL 3rd, Le-Lindqwister N, King D, Rowland KM, Weaver KE, Klepin HD, Shaw EG, Lesser GJ. Phase III Randomized, Placebo-Controlled Clinical Trial of Donepezil for Treatment of Cognitive Impairment in Breast Cancer Survivors After Adjuvant Chemotherapy (WF-97116). J Clin Oncol. 2024 Jul 20;42(21):2546-2557. doi: 10.1200/JCO.23.01100. Epub 2024 May 6. PMID 38709986

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible patients that consented to participate were enrolled and randomized.
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 140 | 136
Completed | 110 | 117
Not Completed | 30 | 19
Not completed — Lost to Follow-up | 5 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Protocol Violation | 6 | 4
Not completed — Too sick or ill | 2 | 1
Not completed — Disease Progression | 1 | 1
Not completed — No reason given | 6 | 4

BASELINE CHARACTERISTICS:
Population: All participants that were enrolled and randomized completed baseline assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 140 | 136 | 276
Age, Customized [Count of Participants; unit: Participants]
  Age: Less than 50 years old | 35 | 35 | 70
  Age: 50-59 years | 52 | 50 | 102
  Age: 60-69 years | 36 | 33 | 69
  Age: 70 years or older | 17 | 18 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 136 | 276
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 5 | 17
  Not Hispanic or Latino | 128 | 131 | 259
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 5 | 11
  White | 128 | 131 | 259
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 140 | 136 | 276
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.9 (6.5) | 31.1 (6.9) | 31.0 (6.7)
Chemotherapy Received [Count of Participants; unit: Participants]
  Anthracycline, cytoxan, and taxane with or without capecitabine | 63 | 63 | 126
  Taxane and cytoxan only | 30 | 31 | 61
  Carboplatin and taxane only | 25 | 26 | 51
  Other combinations | 22 | 16 | 38
Menopausal Status [Count of Participants; unit: Participants] — Participant reported
  Participants
    Perimenopausal or Postmenopausal | 129 | 125 | 254
    Premenopausal | 11 | 11 | 22
Currently taking hormonal therapy [Count of Participants; unit: Participants] — Participant reported use of hormonal therapies (for their breast cancer treatment) at time of study enrollment.
  Participants
    Yes | 95 | 97 | 192
    No | 45 | 39 | 84
Time since completed chemotherapy (months) [Mean (Standard Deviation); unit: months] | 28.8 (14.0) | 30.5 (14.4) | 29.6 (14.2)
Shipley Institute of Living Scale-2 Vocabulary [Mean (Standard Deviation); unit: score on a scale 0-40] — The Shipley Institute of Living Scale-Version 2 Vocabulary subtest was used to estimate premorbid cognitive function (score range, 0-40). Higher values represent better cognitive function.
  score on a scale 0-40 | 30.4 (4.2) | 31.0 (4.2) | 30.7 (4.2)
Highest level of Education Completed [Count of Participants; unit: Participants]
  High School Graduate/GED or less | 28 | 20 | 48
  Some college/vocational training | 55 | 57 | 112
  College degree | 30 | 23 | 53
  Post graduate work or degree | 16 | 21 | 37
  Prefer not to answer or unknown | 11 | 15 | 26
Hopkins Verbal Learning Test- Revised (HVLT-R): Total [Mean (Standard Deviation); unit: score on a scale 0-36] — Hopkins Verbal Learning Test-Revised (HVLT-R): The HVLT-R measures verbal learning and memory. It consists of a 12-item word list which is read to patients on three successive learning trials. Free recall scores are recorded for each learning trial. After a 20-minute interval during which patients complete other non-interfering tasks and questionnaires they are asked to recall the target words. Range is 0-36 with higher values representing better verbal learning and memory.
  score on a scale 0-36 | 23.3 (4.2) | 23.1 (4.7) | 23.3 (4.4)
Hopkins Verbal Learning Test- Revised (HVLT-R): Delayed Recall [Mean (Standard Deviation); unit: score on a scale 0-12] — Measure Description: Hopkins Verbal Learning Test-Revised (HVLT-R): The HVLT-R measures verbal learning and memory. It consists of a 12-item word list which is read to patients on three successive learning trials. Free recall scores are recorded for each learning trial. After a 20-minute interval during which patients complete other non-interfering tasks and questionnaires they are asked to recall the target words. Delayed Recall range is 0-12 with higher values representing better verbal learning and memory.
  score on a scale 0-12 | 8.3 (2.0) | 8.2 (2.1) | 8.3 (2.1)
Hopkins Verbal Learning Test- Revised (HVLT-R): Recognition [Mean (Standard Deviation); unit: score on a scale 0-12] — Measure Description: Hopkins Verbal Learning Test-Revised (HVLT-R): The HVLT-R measures verbal learning and memory. It consists of a 12-item word list which is read to patients on three successive learning trials. Free recall scores are recorded for each learning trial. After a 20-minute interval during which patients complete other non-interfering tasks and questionnaires they are asked to recall the target words. Recognition memory range is 0-12 with higher values representing better verbal learning and memory.
  score on a scale 0-12 | 10.9 (1.2) | 10.9 (1.4) | 10.9 (1.3)
Hopkins Verbal Learning Test- Revised (HVLT-R): Discrimination [Mean (Standard Deviation); unit: score on a scale -12 to 12] — Measure Description: Hopkins Verbal Learning Test-Revised (HVLT-R): The HVLT-R measures verbal learning and memory. It consists of a 12-item word list which is read to patients on three successive learning trials. Free recall scores are recorded for each learning trial. After a 20-minute interval during which patients complete other non-interfering tasks and questionnaires they are asked to recall the target words. Discrimination range is -12 to 12 with higher values representing better verbal learning and memory.
  score on a scale -12 to 12 | 10.3 (1.5) | 10.3 (1.8) | 10.3 (1.6)
Trail Making Test (TMT) - A [Mean (Standard Deviation); unit: seconds] — TMT Part A consists of 25 circles on a piece of paper with the numbers 1 to 25 written randomly in each. For Part A, the person is tasked with drawing a line from one circle to the next in ascending numerical order, from 1 to 25, as quickly as possible. The lines between the circles are referred to as the "trail." Range 1-300 in seconds. Lower values indicate completing task faster with less difficulty. It is a measure of executive functioning with lower values being better.
  seconds | 37.1 (27.1) | 25.8 (23.4) | 36.5 (25.3)
Trail Making Test (TMT) - B [Mean (Standard Deviation); unit: seconds] — TMT Part B also consists of 25 circles on a piece of paper, But, rather than all of the circles containing numbers, they contain numbers (1 to 12) and letters (A through L). For Part B, the person is tasked with connecting the circles in ascending order, alternating back and forth from numbers to letters. In other words, the "trail" would be connected like this:1-A-2-B-3-C-4-D-5-E-6-F-7-G-8-H-9-I-10-J-11-K-12-L-13. The range 1-300 seconds. Higher values indicate worse executive functioning.
  seconds | 91.2 (50.4) | 82.3 (45.7) | 86.9 (48.3)
Controlled Oral Word Association (COWA) [Mean (Standard Deviation); unit: score on scale 0 to no specified maximum] — The Controlled Oral Word Association Test from the Halstead-Reitan Neuropsychological Battery is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe (typically 60 seconds). Scores are the sum of all acceptable words. Minimum is 0 with no specified maximum; higher values represent better verbal fluency.
  score on scale 0 to no specified maximum | 34.7 (10.1) | 34.8 (10.3) | 34.7 (10.2)
Digit Span Test Backward [Mean (Standard Deviation); unit: score on a scale 0-16] — The Digit Span Task (Backwards-Only Child Version) measures working memory. On each question the participant repeats the numbers in reverse order of that presented aloud by the examiner (e.g., If the examiner says "5-6", the correct response would be "6-5"; If the examiner says "5-1-7-4-2-3-8", the correct response would be "8-3-2-4-7-1-5"). Score is 0 to 16 with higher scores representing better working memory.
  score on a scale 0-16 | 6.4 (2.2) | 6.8 (2.2) | 6.5 (2.2)
Digit Symbol Coding [Mean (Standard Deviation); unit: scores on a scale 0-100] — The digit symbol test measures processing speed, working memory, visuospatial processing, and attention. Scores range from 0 to 100, with higher scores indicating higher cognitive function.
  scores on a scale 0-100 | 64.2 (17.3) | 61.6 (16.5) | 62.9 (17.0)
The Functional Assessment of Cancer Therapy (FACT)-Cognition: Perceived Cognitive Impairment [Mean (Standard Deviation); unit: scores on a scale 0-80] — The Functional Assessment of Cancer Therapy (FACT)-Cognition is a patient-reported outcome (PRO) that includes subscales to measure Perceived Cognitive Impairment (PCI, n = 20 items, score range 0-80). Higher FACT-Cog PCI scores are better and indicate less cognitive impairment.
  scores on a scale 0-80 | 29.2 (14.8) | 33.4 (15.9) | 31.3 (15.5)
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue - Short Form 7a [Mean (Standard Deviation); unit: T-score] — This self-report scale assesses fatigue. Scores range from 7 to 35 and are converted to a T-scale with ranges from 29.4 to 83.2. Higher scores representing more fatigue.
  T-score | 55.5 (7.8) | 55.4 (8.0) | 55.5 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) - Total
Description: Hopkins Verbal Learning Test-Revised (HVLT-R): The HVLT-R measures verbal learning and memory. It consists of a 12-item word list which is read to patients on three successive learning trials. Free recall scores are recorded for each learning trial. After a 20-minute interval during which patients complete other non-interfering tasks and questionnaires they are asked to recall the target words. Range is 0-36 with higher values representing better verbal learning and memory.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat analysis. Considered and utilized all data available at each timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale of 0-36
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
score on a scale of 0-36
  12 Weeks | 24.4 [23.6 to 25.1] | 24.5 [23.7 to 25.3]
  24 Weeks | 26.0 [25.2 to 26.8] | 26.5 [25.8 to 27.2]
  36 Weeks | 25.1 [24.3 to 25.9] | 25.9 [25.1 to 26.7]
Statistical Analysis 1: Comparison: Donepezil vs Placebo; With a sample size of 266, there was 90% power to detect a treatment difference of 2 words for HVLT-R total recall score (SD=4.26, effect size=0.47) with a two-sided 5% level of significance. This calculation assumed an ANCOVA model analysis with 25% dropout and 2% missing data at end of treatment. A single interim analysis for futility occurred after 138 participants, with stopping rule of two-sided p-value < 0.0154. This design required 3.5% more than fixed design, increasing total to 276; Test type: Superiority — Mixed effects repeated measures analysis of covariance (RMANCOVA) models with covariates of treatment, time, time by treatment interaction, baseline outcome level, age stratification and an unstructured covariance matrix. The primary objective was assessed using a linear contrast of group effect at 24 weeks; p = 0.32, ANCOVA

2. Secondary Outcome: Digit Symbol Coding Results
Description: The digit symbol coding (DSC) test measures processing speed, working memory, visuospatial processing, and attention. The DSC test measures processing speed. It requires respondents to transcribe symbols (e.g., >) associated with a number (0-9) into empty boxes beneath a series of randomly ordered numbers. Total score is number of correctly transcribed symbols in 2 minutes. Scores range from 0 to 100, with higher scores indicating higher cognitive function.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat analysis. All available data from all participants utilized in models.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 0-100
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
score on a scale 0-100
  12 Weeks | 69.6 [67.1 to 72.1] | 67.7 [65.2 to 70.2]
  24 Weeks | 71.9 [69.4 to 74.5] | 71.9 [69.4 to 74.4]
  36 Weeks | 74.2 [71.4 to 76.9] | 71.7 [69.1 to 74.3]

3. Secondary Outcome: PROMIS 7-item Fatigue Scale Converted to T-scale Results
Description: This self-report scale assesses fatigue. Scale ranges from 7 to 35 converted to T-scale ranging 29.4 to 83.2 Higher scores representing more fatigue.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat: all participants and timepoints available were utilized.
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
T-score
  12 Weeks | 52.3 [51.2 to 53.5] | 53.0 [51.8 to 54.1]
  24 Weeks | 51.8 [50.6 to 53.0] | 52.0 [50.9 to 53.2]
  36 Weeks | 52.2 [51.0 to 53.3] | 53.0 [51.9 to 54.1]

4. Secondary Outcome: FACT-Cognition (Version 3): Perceived Cognitive Impairment
Description: The FACT-Cog is a patient-reported outcome (PRO) that includes subscales to measure Perceived Cognitive Impairment (PCI, n = 20 items, score range 0-80). Higher FACT-Cog PCI scores are better and indicate less cognitive impairment.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat analyses: all available timepoints and participant data utilized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 0-80
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
score on a scale 0-80
  12 Weeks | 45.6 [43.0 to 48.1] | 45.6 [43.1 to 48.1]
  24 Weeks | 49.4 [46.7 to 52.1] | 48.8 [46.1 to 51.4]
  36 Weeks | 47.6 [45.0 to 50.3] | 47.5 [44.9 to 50.0]

5. Secondary Outcome: Controlled Oral Word Association Test (COWA) Results
Description: The Controlled Oral Word Association Test from the Halstead-Reitan Neuropsychological Battery is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe (typically 60 seconds). Scores are the sum of all acceptable words. Minimum is 0 with no specified maximum; higher values represent better verbal fluency.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat analysis. All available timepoints from all participants utilized.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 0 to no specified maxim
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
score on a scale 0 to no specified maxim
  12 Weeks | 6.7 [6.3 to 7.1] | 6.6 [6.2 to 7.0]
  24 Weeks | 6.9 [6.4 to 7.3] | 7.0 [6.6 to 7.4]
  36 Weeks | 6.8 [6.3 to 7.2] | 7.3 [6.8 to 7.7]

6. Secondary Outcome: Trail Making Test, Parts A & B (TMT-A, TMT-B) Results
Description: TMT Part A consists of 25 circles on a piece of paper with the numbers 1 to 25 written randomly in each. For Part A, the person is tasked with drawing a line from one circle to the next in ascending numerical order, from 1 to 25, as quickly as possible. The lines between the circles are referred to as the "trail." Range 1-300 in seconds. Lower values indicate completing task faster with less difficulty. It is a measure of executive functioning with lower values being better.
  TMT Part B also consists of 25 circles on a piece of paper, But, rather than all of the circles containing numbers, they contain numbers (1 to 12) and letters (A through L). For Part B, the person is tasked with connecting the circles in ascending order, alternating back and forth from numbers to letters. In other words, the "trail" would be connected like this:1-A-2-B-3-C-4-D-5-E-6-F-7-G-8-H-9-I-10-J-11-K-12-L-13. The range 1-300 seconds. Higher values indicate worse executive functioning.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat analysis. All available participants and time points utilized.
Measure: Least Squares Mean (95% Confidence Interval); unit: time (seconds)
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
time (seconds)
  TMT-A 12 Weeks | 32.8 [28.6 to 36.9] | 34.1 [30.0 to 38.1]
  TMT-A 24 Weeks | 31.4 [28.6 to 34.3] | 29.9 [27.1 to 32.7]
  TMT-A 36 Weeks | 28.8 [26.3 to 31.4] | 30.4 [28.0 to 32.8]
  TMT-B 12 Weeks | 76.7 [70.7 to 82.7] | 78.1 [72.3 to 83.9]
  TMT-B 24 Weeks | 74.8 [68.6 to 80.9] | 75.1 [69.2 to 81.1]
  TMT-B 36 Weeks | 70.1 [65.2 to 75.0] | 73.6 [68.9 to 78.2]

7. Secondary Outcome: Digit Span Test-Backwards (DST-B)
Description: The Digit Span Task (Backwards-Only Version) measures working memory. On each question the participant repeats the numbers in reverse order of that presented aloud by the examiner (e.g., If the examiner says "5-6", the correct response would be "6-5"; If the examiner says "5-1-7-4-2-3-8", the correct response would be "8-3-2-4-7-1-5"). Score is 0 to 16 with higher scores representing better working memory.
Time Frame: Baseline, Weeks 12, 24, 36
Population: Intent to treat analyses: all timepoints and participant data used.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale 0-16
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 140 | 136
score on a scale 0-16
  12 Weeks | 6.7 [6.3 to 7.1] | 6.6 [6.2 to 7.0]
  24 Weeks | 6.9 [6.4 to 7.3] | 7.0 [6.6 to 7.4]
  36 Weeks | 6.8 [6.3 to 7.2] | 7.3 [6.8 to 7.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline, 3 weeks, 6 weeks, 12 weeks, 24 weeks, and 36 weeks. And participants could report additional events at any time.
Description: Each adverse event will include the date of onset, date of resolution, severity, and the relationship to the study agent or intervention, and any action taken with respect to the study agent or intervention. Grade 1 and 2 adverse events (AEs), expected grade 3 or grade 4 AEs will not be collected. Unexpected grade 3 AEs that are unrelated or unlikely will also not be collected.
Arm/Group | Donepezil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/136
Serious Adverse Events (participants affected / at risk) | 12/140 | 8/136
Other Adverse Events (participants affected / at risk) | 0/140 | 0/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=140) | Placebo (N=136)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain (Investigations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Weight Gain (Investigations) | 0 (0) | 1 (1)
Constitutional Symptoms Other (Investigations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Our mainly non-Hispanic, white sample of breast cancer survivors, while geographically diverse, is not representative of all survivors. A lack of validated alternate forms of most of our tests may have contributed to a practice effect. We did not collect estrogen receptor, progesterone receptor or human epidermal growth factor receptor 2 (HER2) status.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT02822573/Prot_SAP_001.pdf
  • Informed Consent Form (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT02822573/ICF_000.pdf